CLINICAL TRIAL: NCT05587270
Title: CLIMB: Climbers' Longitudinal Attitudes to Injuries, Mental Health and Body Image
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Sophiahemmet University (Other)
Responsible Party: Sponsor
Other Study IDs: CLIMB
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Mental Health Issue; Musculoskeletal Pain; Eating Disorders; Relative Energy Deficiency in Sport
Keywords: Depression; Anxiety; Stress; Pain; Rock climbing; Eating disorders; Cohort
MeSH Terms: conditions — Musculoskeletal Pain; Feeding and Eating Disorders; Relative Energy Deficiency in Sport; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rock Climbers: The whole eligible population of Swedish climbers on elite- or sub-elite levels of competition will be invited to participate in the study. Participants will be both male and female, 13 years and older. There are approximately 40 climbers eligible at elite level and a minimum of 80 climbers at sub-elite level of competition.
  Interventions: Other: Web based surveys; Radiation: DXA
- Controls: A non-athlete control group (n matched to the study group) from the general population, will be invited to participate in the study.
  Interventions: Other: Web based surveys

INTERVENTIONS:
Other: Web based surveys — A web-based survey will explain the purpose, aims, and ethical rights, as well as how to complete the questionnaire online. Further, information about, and an invitation to participate in the DXA-scan will be included with this information. Upon electronic consent by both parent and athlete (or just athlete if of consenting age (15 y o a)), access to the multi-section questionnaire will be granted. Contact details of the researchers will be available in case of difficulties comprehending the questions. Following completion, the participants' data will be sent to a secure database for analysis. Participants will be ensured of the confidentiality of the study and will be free to withdraw from the study. Parents will also be asked to provide their consent if participants age is under 14.
Radiation: DXA — All participants will be invited to complete a DXA scan at baseline. DXA is to date the most reliable way of examining the long-term physical consequences of RED-S.
  Groups: Rock Climbers

SUMMARY:
Eating disorders (ED) are serious mental illnesses with high mortality rates and significant impact on an individual's quality of life. These disorders are characterized by preoccupation of weight and shape, leading to restrictive eating behavior and compensatory behaviors (purging and excessive/compulsive exercise). Comorbidities with mental health problems are common. Athletes in leanness-focused sports report higher levels of EDs compared to athletes from sports without such focus . Energy Availability (EA) has been suggested the key variable in "Relative Energy Deficiency in Sports" (RED-S) with studies reporting impairment of reproductive function and bone formation.

Climbing is a weight sensitive sport where athletes generally, benefit from a lean body shape and low weight, a risk factors for ED. Therefore, climbing athletes can be expected to be at high-risk to develop these conditions. To our knowledge, there are no studies on the prevalence and magnitude of EDs among climbers. Due to the overrepresentation of EDs reported in sports and the poor treatment prognosis, early detection and prevention of ED symptoms are essential. The present study will study the prevalence of ED symptoms, changes over time and trajectories of key variables along with related problem areas such as bone health and mental health problems in order to take steps towards tailored strategies for the prevention of EDs in climbing.

The overall purpose of the project is to study prevalence and changes over a two-year period (with a planned follow-up period of up to five years) of eating disordered (ED) symptoms, mental health problems, overuse injuries, bone health as well as indications of relative energy deficiency (RED-S) in elite vs. sub-elite Swedish climbers. Climbers will be compared to a group of normal controls. Further, differences will be studied in groups with high vs. low levels of EDs, comparing occurrence of mental health problems, overuse injuries and bone health. Trajectories of mentioned variables over time will be analyzed.

DETAILED DESCRIPTION:
Study objectives:

The overall purpose of the project is to study prevalence and changes over a two-year period (with a planned follow-up period of up to five years) of eating disordered (ED) symptoms, mental health problems, overuse injuries, bone health as well as indications of relative energy deficiency (RED-S) in elite and sub-elite Swedish climbers. Climbers will be compared to a group of normal controls. Further, differences will be studied in groups with high vs. low levels of EDs, comparing occurrence of mental health problems, overuse injuries and bone health. Trajectories of mentioned variables (with the exception of bone health) over time will be analyzed.

Specific research questions:

A) BASELINE

To determine the prevalence of disordered eating behaviors, mental health problems, compulsive training, self-reported symptoms of LEA, overuse injuries and bone density in advanced to elite climbers compared to controls.

Are there gender differences among climbing athletes as far as ED symptoms, body image, compulsive training, perfectionism, mental health problems, sleep quality and overuse injuries?

Do climbing athletes at higher levels of competition (elite vs. advanced) report differing levels of symptoms related to disordered eating behaviors, mental health problems, compulsive training, self- reported symptoms of LEA, overuse injuries and bone density than normal controls?

Are there difference between climbing athletes reporting differences in ED symptoms respectively with regards to bone health as measured by Dual-Energy X-ray Absorptiometry (DXA).

B) FOLLOW UP

To study the trajectories of mentioned variables over time and examine the association between modifiable risk factors and ill health and outcome measured by DASS21, EDEQ and OSLO SPORTS OVERUSE INJURIES QUESTIONNAIRE.

Study design:

The study design is longitudinal using a web-based questionnaire with four measures over a two-year period (baseline, 6-, 12- and 24 months) and additional follow-ups at 3 and 5 years after baseline. The whole eligible population of Swedish climbers on elite- or sub-elite levels of competition will be invited to participate in the study. Participants will be both male and female, 13 years and older. There is a minimum of 40 climbers eligible at elite level and a minimum of 80 climbers at sub-elite level of competition. A non-elite athlete control group (n matched of the climbing group) from the general population, will be invited to participate in the study.

In addition to the web-based questionnaire, participants will be invited to the measurement of bone health using DXA at the baseline measurement.

Source population:

The whole eligible population of Swedish climbers on elite- or sub-elite levels of competition will be invited to participate in the study. Participants will be both male and female, 13 years and older.

Sample size: To our knowledge, no previous research has been presented and since the climbing population is small, and the expected outcome measures (ED-symptoms, mental health problems, injuries and bone health) are unknown, we will not be able to carry out power calculations. However, based on similar injury research by one of the co-applicants, a power calculation was estimated on standard deviation of 1.0, significant level set to 0.05, and statistical power 0.80. The study needed 38 participants in each group to detect estimated group differences. We will therefore include at least 40 in each group.

Data collection

The study has been endorsed by the Swedish Climbing Federation. Study information will be distributed via the federation to national teams and clubs asking them to distribute the web-based survey link (computed by the research team) to the climbing athletes and controls. The web-based survey will explain the purpose, aims, and ethical rights, as well as how to complete the questionnaire. Further, information regarding, and an invitation to participate the DXA-scan will be included with this information. Upon electronic consent by both parent and athlete (or just athlete if of consenting age (15 y o a)), access to the multi-section questionnaire will be granted. Contact details of the researchers will be available in case of difficulties comprehending the questions. Following completion, the participants' data will be stored at a secure database for analysis. Participants will be ensured of the confidentiality of the study and will be free to withdraw from the study at any time. Appointments for DXA-scans will be set up after informed consent has been established for the study as a whole.

Exposures

Rock-climbing

Outcomes

Eating Disorders: The Eating Disorders Questionnaire (EDE-Q 6.0) will be used and consists of four subscales: restraint, eating concern, shape concern and weight concern, addressing core dimensions of eating disorders (Berg et al., 2012).

Overuse injuries: The Oslo Sports Trauma Research Center Overuse Injury Questionnaire (OSTRC-O; Clarsen et al., 2020) will be used and measures athlete's self-reported a) participation in sport, b) modified training/competing,c) performance and d) pain in a 4-grades scale from full participation to could not participate due to problems (of injury).

Perfectionism: The Frost Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart & Rosenblate, 1990) will be used, utilizing the subscales of personal standards (PS) and concern over mistakes (CM).

Compulsive Exercise: Weight loss behaviors and emotion regulation using training is measured with Compulsive Exercise Test (CET; Taranis, Touyz & Meyer, 2011). The subscales included are: "Weight control exercise" (WCE) and "Avoidance of negative affect and rule driven behavior" (ANARDB).

Body Image: The brief version of the 8 item Body Shape Questionnaire, (BSQ-8C; Welch, Lagerström & Ghaderi, 2012) will be used.

Symptoms of mental health problems are measured by the Depression Anxiety Stress Scale (DASS-21; Lovibond & Lovibond, 1995).

Sleep quality: The Pittsburg Sleep Quality Index (PSQI; Carpenter & Andrykowski,1998) will be used and includes 19 items addressing seven subscales: sleep duration, efficiency, quality, latency, medication use, disturbances and daytime dysfunctions.

Basic symptoms indicative of RED-S will be assessed by 17 questions about meal pattern, menstrual function and injuries. These questions were developed and previously used with a Swedish figure skating population, 13 years and older (n=224; Edlund, 2020).

Dual-Energy X-ray Absorptiometry (DEXA) will be carried out on both athletes and controls, comparing bone mineral density between the groups at baseline.

Data analysis and statistics:

Group comparisons between climbers and controls examining the difference between the above-mentioned variables between the study groups. Specific tests will be depending on the type of data, distribution of the variables and the size of the study population.

Group comparisons examining gender differences among climbers regarding the above-mentioned variables. Specific tests will be depending on the type of data, distribution of the variables and the size of the study population.

Group comparisons examining differences among climbers of different level (Elite and advanced) regarding the above-mentioned variables. Specific tests will be depending on the type of data, distribution of the variables and the size of the study population.

Associations in climbers between ED symptoms with regards to bone health as measured by Dual-Energy X-ray Absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

* Age over 13

Specific inclusion criteria for the study group:

* Men: completed a boulder route rated harder than 6b or a lead route rated 7a+ within the last three months.
* Women: completed a boulder route rated harder than 6a or a lead route rated 6c within the last year.

Exclusion Criteria for the study group:

* None

Exclusion criteria for the control group:

* Previous or current participation on elite level in any sport.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All individuals invited to participate in the study will answer the question about sex (female or male). All analysis with regard to sex in the study are based on these categories.
Study Population: The whole eligible population of Swedish climbers on elite- or sub-elite levels of competition will be invited to participate in the study. Participants will be both male and female, 13 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 366 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Eating disorders | 2022-2025
  Eating Disorders: The Eating Disorders Examination-Questionnaire (EDE-Q 6.0) will be used and consists of four subscales: restraint, eating concern, shape concern and weight concern, addressing core dimensions of eating disorders (Berg et al., 2012). Higher scores on the global scale and subscales denote more problematic eating behaviours and attitudes. A cut-off of 2 on the global scale indicate a sublclinical eating disorder and a score of 4 or higher on the global score is generally used as clinically significant.
Relative energy deficiency | 2022-2025
  Basic symptoms indicative of RED-S will be assessed by 17 questions about meal pattern, menstrual function and injuries. These questions were developed and previously used with a Swedish figure skating population, 13 years and older (n=224; Edlund, 2020).

SECONDARY OUTCOMES:
Sleep quality | 2022-2025
  The Pittsburg Sleep Quality Index (PSQI; Carpenter & Andrykowski,1998) will be used and includes 19 items addressing seven subscales: sleep duration, efficiency, quality, latency, medication use, disturbances and daytime dysfunctions. In scoring the PSQI, the seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Depression, anxiety and stress | 2022-2025
  Symptoms of mental health problems are measured by the Depression Anxiety Stress Scale (DASS-21; Lovibond & Lovibond, 1995).
  The outcome is nominal with categories according to the following:
  Depression:
  Normal 0-9 Mild 10-12 Moderate 13-20 Severe 21-27 Extremely severe 28-42.
  Anxiety:
  Normal 0-6 Mild 7-9 Moderate 10-14 Severe 15-19 Extremely severe 20-42.
  Stress:
  Normal 0-9 Mild 10-12 Moderate 13-20 Severe 21-27.
Body Image | 2022-2025
  The brief version of the 8 item Body Shape Questionnaire, (BSQ-8C; Welch, Lagerström & Ghaderi, 2012) will be used. The outcome is nominal with categories according to the following:
  No concern with shape <19. Mild concern with shape 19-25. Moderate concern with shape 26-33. Marked concerns with shape >33)
Compulsive Exercise | 2022-2025
  Weight loss behaviors and emotion regulation using training is measured with Compulsive Exercise Test (CET; Taranis, Touyz & Meyer, 2011). The subscales included are: "Weight control exercise" (WCE) and "Avoidance of negative affect and rule driven behavior" (ANARDB). The CET is a self-reported questionnaire designed to explore the emotional, cognitive and behavioral characteristics of compulsive exercise. It comprises 24 items answered on a 6-point Likert scale, from 0 (never true) to 5 (always true). CET consists of five subscales: "avoidance and rule-driven behavior," "weight control exercise," "mood improvement," "lack of exercise enjoyment," and "exercise rigidity." Mean scores of each subscale are measured.
Perfectionism | 2022-2025
  The Frost Multidimensional Perfectionism Scale (FMPS; Frost, Marten, Lahart & Rosenblate, 1990) will be used, utilizing the subscales of personal standards (PS) and concern over mistakes (CM). The outcome is dichotomous with a cut off score of >29.
Overuse injuries | 2022-2025
  The Oslo Sports Trauma Research Center Overuse Injury Questionnaire (OSTRC-O; Clarsen et al., 2020) will be used and measures athlete's self-reported a) participation in sport, b) modified training/competing,c) performance and d) pain in a 4-grades scale from full participation to could not participate due to problems (of injury).

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sansone, M.D, Ph.D., Principal Investigator — Göteborg University
Locations (1):
- Göteborg University, Gothenburg, Västergötaland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Parallel studies are in planning with Universities of Norway for cross-cultural comparisons with merged data sets.

REFERENCES:
- [Derived] Nigicser I, Identeg F, Sansone M, Hedelin H, Forsberg N, Tranaeus U, Edlund K. Do Swedish rock-climbers exhibit more eating disorder and body dissatisfaction symptoms than non-climbers? A cross-sectional study. BMJ Open. 2024 Oct 16;14(10):e085265. doi: 10.1136/bmjopen-2024-085265. PMID 39414282
- [Derived] Edlund K, Nigicser I, Sansone M, Identeg F, Hedelin H, Forsberg N, Tranaeus U. Protocol for a 2-year longitudinal study of eating disturbances, mental health problems and overuse injuries in rock climbers (CLIMB). BMJ Open. 2023 Sep 13;13(9):e074631. doi: 10.1136/bmjopen-2023-074631. PMID 37709336